CLINICAL TRIAL: NCT07188597
Title: Culturally Adapted Cognitive Behavior Therapy for Individuals At Risk of First Episode Psychosis: A Mixed Method Study
Brief Title: Culturally Adapted Cognitive Behavior Therapy for Individuals At Risk of First Episode Psychosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PILL-CBT ARMS-FEP
Record Dates: First submitted 2025-09-16; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Individuals at Risk of First Episode Psychosis
MeSH Terms: interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Cognitive Behavior Therapy for those at risk of first episode psychosis- "evidence-based therapy for people with ARMS" (Van der Gaag, et al., 2013).
  The participants in the intervention group will receive a culturally adapted manualised cognitive behavioral therapy (CBT). The interventions aim to reduce symptoms, normalises psychosis-like experiences and prevents a catastrophic appraisal of the psychotic-like symptoms from occurring.
Who Masked: Outcomes Assessor
Masking Description: Researchers conducting outcome assessments will be blind to treatment allocations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Behavior Therapy for those at risk of first episode psychosis (Experimental): The participants in the intervention group will receive a culturally adapted manualised cognitive behavioral therapy (CBT). The interventions aim to reduce symptoms, normalises psychosis-like experiences and prevents a catastrophic appraisal of the psychotic-like symptoms from occurring
  Interventions: Behavioral: Cognitive Behavior Therapy for those at risk of first episode psychosis
- Treatment as Usual (No Intervention): Treatment As Usual (TAU):
  Local medical, psychiatric and primary care services provide standard routine care according to their clinical judgment and available resources. These participants will receive an initial assessment along with TAU as ascertained by their treating doctor at the hospital. In current practice, individuals with ARMS (at risk of first episode psychosis) are not routinely referred to any psychological service in Pakistan. TAU in Pakistan largely comprises of pharmacotherapy. Research staff will record the nature and intensity of the routine care delivered for each participant.

INTERVENTIONS:
Behavioral: Cognitive Behavior Therapy for those at risk of first episode psychosis — Participants will receive a culturally adapted manualised Cognitive Behavioural Therapy (CBT) for those at risk of first episode psychosis (FEP). The intervention aims to reduce symptoms, normalise psychosis-like experiences, and prevent catastrophic appraisals that may lead to delusions. It integrates psychoeducation, behavioural experiments, and techniques addressing cognitive biases. By reframing unusual experiences as perceptual or reasoning biases, distress and emotional arousal are reduced, lowering the chance of fixed, frightening beliefs. Homework tasks further support coping. CBT for At-Risk Mental States has shown effectiveness in reducing transition to psychosis and improving recovery. This study will adapt and field test the manual, with potential for remote delivery via phone, video, or AI tools to enhance accessibility.
  Other Names: CBT-FEP
  Arms: Cognitive Behavior Therapy for those at risk of first episode psychosis

SUMMARY:
Young people constitute nearly half of Pakistan's population and are highly vulnerable to risk factors for mental illness, including poverty, inequality, abuse, and violence. Estimates suggest that 19-34% of children and adolescents experience emotional or behavioural disorders, though this is likely underestimated. In recent years, research has focused on those at imminent risk of developing serious conditions such as first episode psychosis. The concept of an At-Risk Mental State (ARMS) has highlighted the urgent need for interventions that address current symptoms, improve functioning, and reduce transition to psychosis.

Up to 80% of young people with ARMS have another diagnosable condition, and almost half show poor psychosocial outcomes even six years after initial help-seeking. Evidence demonstrates that early identification and treatment can delay or prevent psychosis, including severe and enduring illnesses like schizophrenia. Cognitive Behaviour Therapy (CBT) is among the most effective evidence-based approaches for this group. However, existing evidence comes largely from high-income countries, raising concerns about cultural applicability in low-resource settings.

This study will culturally adapt and field test a manualised CBT intervention for young people at risk of first episode psychosis. To our knowledge, this is the first such study in a low-income country. Findings will inform scalable, culturally relevant interventions for Pakistan and similar contexts.

DETAILED DESCRIPTION:
Aims and Objectives:

The study has following aims and objectives:

1. To culturally adapt the existing Cognitive Behavior Therapy for those at risk of first episode psychosis- "evidence-based therapy for people with ARMS" (Van der Gaag, et al., 2013).
2. To field test the culturally adapted intervention in a randomised controlled trial
3. To check whether adapted intervention reduces or delay the rates or incidence of transition from ARMS to first episode psychosis;
4. To check whether adapted intervention improves other symptoms such as depression, anxiety and/or level of functioning in ARMS
5. To explore the pereceived usefulness of intervention including perceived barriers and facilitators from different stakeholders' perspective.

Feasibility and acceptability of the intervention is defined as:

* Recruitment rates, attendance (attending more than 70% of intervention sessions)
* Acceptability of the intervention (based on participants satisfaction, attendance, attrition rates)
* Completeness of assessment tools and the assessment schedule by participants

  * Preliminary efficacy of the intervention

ELIGIBILITY:
Inclusion Criteria:

* Male or female help-seeking individual aged 16-35 years;
* Score 6 or above on PQ-16
* Meet the at risk of FEP criteria using CAARMS Operationalized Intake Criteria based on three groups (vulnerability, attenuated psychosis or brief limited intermittent psychotic symptoms group);
* Assessed as competent to provide informed consent.
* Give written informed consent.

Exclusion Criteria:

* Temporary resident unlikely to be available for follow up.
* Unable to engage, participate or respond to research questionnaires.
* a history of psychotic illness (treated or untreated).
* previous treatment with an antipsychotic or mood-stabilising agent.
* active substance abuse (except nicotine or caffeine) or dependence within the last three months, according to DSM-V criteria.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility Indicator | From baseline to 12th week (end of intervention)
  feasibility will be determined by collecting data on recruitment and retention rates, The success criterion of feasibility will be to recruit > 50% of eligible participants
Acceptability Indicator | From baseline to 12th week (end of intervention)
  Intervention acceptability will be assessed using data on attendance. Criterion for acceptability is a mean attendance rate of >70%.

OTHER OUTCOMES:
The Prodromal Questionnaire | From baseline to 12th week (end of intervention)
  A brief 16-item self-report screening questionnaire assesses the presence of attenuated psychotic symptoms on a two-point scale (true/false) followed by a 4-point distress rating for each item. A cut of 6 or above considered for further assessment to confirm at risk criteria
Brief-Comprehensive Assessment of At-Risk Mental States | From baseline to 12th week (end of intervention)
  A semi-structured interview that assists in the identification of individuals at risk of developing a first-episode psychotic disorder.
Client Satisfaction Questionnaire | From baseline to 12th week (end of intervention)
  The participants will rate their satisfaction with treatment at 3 months (after completion of the intervention) using the CSQ
Calgary Depression Scale | From baseline to 12th week (end of intervention)
  The Calgary Depression Scale for Schizophrenia (CDSS) is a depression rating scale especially developed for assessing depression in schizophrenia. Higher score shows higher depression
Health Related Quality of Life EQ-5D-5L | From baseline to 12th week (end of intervention)
  The EQ-5D is a generic instrument for describing and valuing health. It is based on a descriptive system that defines health in terms of 5 dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension has 5 response categories corresponding to no problems, some problems, and extreme problems
Generalized Anxiety Disorder (GAD-7) | From baseline to 12th week (end of intervention)
  GAD-7 is a brief scale to identify probable cases of generalised anxiety and depression, as well as assessing symptom severity. Higher scores shows greator severity of anxiety
Social and Occupational Functioning Scale (SOFAS) | From baseline to 12th week (end of intervention)
  SOFAS will be used to assess overall functioning in a single score (0-100). It is a global rating of current functioning; this instrument focuses on social and occupational functioning that is independent of the overall severity of the individual's psychological symptoms.
Brief Illness Perception Questionnaire | From baseline to 12th week (end of intervention)
  a nine-item scale designed to rapidly assess the cognitive and emotional representations of illness
Kessler Psychological Distress Scale | From baseline to 12th week (end of intervention)
  Level of distress will be assessed using a 10-item scale the "Kessler Psychological Distress Scale

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Commuity/Schools/Colleges, Karachi, Sindh
  - Karwan e Hayat, Karachi, Sindh